CLINICAL TRIAL: NCT00305266
Title: "Clinical Study of Intravenous Immunoglobulin Treatment of Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy"
Brief Title: Study of CIDP Patients During IVIG Treatment
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Other Study IDs: 2005-0018; EudraCT nr.: 2004-004357-26
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2007-11

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
Keywords: CIDP; IVIG; gammaglobulin; Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: intravenous gammaglobulin — individual dose

SUMMARY:
The aim of this study is to quantify the effect of IVIG treatment in a group of patients with chronic inflammatory demyelinating polyradiculoneuropathy(CIDP), who requires continues treatment of IVIG at regular intervals of 3-10 weeks:

1. During continues treatment of IVIG at regular intervals of 3-10 weeks.
2. During pause in treatment.

Hypothesis:

1. The disease activity in the patients are cyclical correlating to the treatment intervals.
2. Pause in treatment will increase disease activity, which can be quantified with symptom scores, disability scales, and clinical test.

Primary effect parameter is muscle strength quantified by isokinetic dynamometry.

Added to the protocol there is an immunological study of inflammatory markers in blood samples of patients under treatment pause.

DETAILED DESCRIPTION:
Background: Chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) is a rare autoimmune disease of the peripheral nervous system characterized by demyelination of the nerves, which causes muscle weakness and sensory loss. Treatment is immune modulating, and intravenous immunoglobulin (IVIG) is first line therapy.Several trials have demonstrated effect on motor function by the initial treatment, but the effect of consecutive IVIG treatment is only sporadic described in the literature.

It is a clinical study including present CIDP patients in treatment at the University Hospital of Aarhus. The patients will be evaluated several times before and after IVIG treatment, to describe the effect profile.

The primary effect parameter is muscle strength quantified by isokinetic dynamometry at ankle knee, hip, wrist, elbow and shoulder. That is a sensitive method of measuring the strength of the larger muscle groups, correlating with symptoms and signs of neuropathy.

Severity of neuropathy among the patients will also be described applying nerve conduction studies, quantitative sensory testing of threshold for detecting vibration and cold at upper and lower limbs, the Neuropathy Disability Scale, the Neuropathy Symptom Score,the overall disability sum score, 9 hole peg test, walking test, and the Short-form 36 health questionnaire.

Added to the protocol there is an immunological study of inflammatory markers in blood samples of patients under treatment pause.

Objective:

With this study we will describe some important aspects in the immune response causing the inflammatory lesions in CIDP and MMN, including:

1. Recruitment of immune cells to the affected tissue by chemoattraction. (Chemokine receptors on mononuclear cells)
2. Crossing the blood-nerve barrier: interactions and adhesion between the lymphocyte and endothelial cell, transendothelial diapedesis and enzymatic degeneration of the basal lamina.(Adhesion molecules on mononuclear cells and soluble in plasma, metalloproteinases)
3. Synthesis of mRNA and secretion of regulatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Motor and sensory dysfunction involving more than one limb.
* Electrodiagnostic study with signs of demyelination

Exclusion Criteria:

* Prior systemic allergic reaction to IVIG
* Severe systemic disease
* Other conditions associated with neuropathy (eg diabetes, lack of vitamin- B12)
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-08; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, MD, Principal Investigator — Aarhus University Hospital; Johannes Jakobsen, professor, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Neurology, Aarhus, Denmark